CLINICAL TRIAL: NCT02906527
Title: Benefit/Risk in Real Life of New Oral Anticoagulants and Vitamin K Antagonists in Patients Aged 75 Years and Over Suffering From Non Valvular Atrial Fibrillation (nv AF) : An Observational Study Conducted on the French Health Insurance Database (SNIIRAM)
Brief Title: Benefit/Risk in Real Life of New Oral Anticoagulants and Vitamin K Antagonists in Patients Aged 75 Years and Over Suffering From Non Valvular Atrial Fibrillation (nv AF)
Acronym: Presage-Aco
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 16DBT-Presage-Aco
Record Dates: First submitted 2016-09-07; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Non Valvular Atrial Fibrillation (nv AF)
Keywords: Cardiology; Oral anticoagulants; Risk and Benefit analysis; Health insurance databases; Safety; Elderly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-exposed group: Non-exposed group / Patients receiving VKA
  Interventions: Drug: Non-exposed group
- Exposed group: Exposed group / Patients receiving DOAC
  Interventions: Drug: Exposed group

INTERVENTIONS:
Drug: Non-exposed group — Non-exposed group / Patients receiving VKA
  Other Names: Patients receiving VKA
  Groups: Non-exposed group
Drug: Exposed group — Exposed group / Patients receiving DOAC
  Other Names: Patients receiving DOAC
  Groups: Exposed group

SUMMARY:
"The aim of the study is to compare, in real life, the risk benefit (including both major bleeding and thrombotic events (TE) and death from any cause) associated with direct oral anticoagulants (DOAC) and with anti vitamin K (VKA) in older adults (≥ 75 years) suffering from nvAF.

The study will be conducted in the French Health insurance database (SNIIRAM). Data of octo+ patients newly treated with an oral anticoagulant (VKA or DOAC) for non valvular atrial fibrillation (nv AF) will be collected from the first exposure of the patient to the drug of interest during the inclusion period to the end of the follow-up period (at least one year of follow-up for each patient)."

DETAILED DESCRIPTION:
"• Context: Oral anticoagulation is recommended for prevention of stroke and thrombo-embolic events in people aged 80 years and over (octo+) suffering from non valvular atrial fibrillation (nv AF) and without contraindication to anticoagulant therapy. Two drug classes are available to achieve this oral anticoagulation: the vitamin K antagonists (VKA, warfarin, fluinione and acenocoumarol) or the Direct Oral Anticoagulants (DOAC, dabigatran, rivaroxaban and apixaban). The data of evidence-based and post-marketing literature on the benefit/risk ratio of DOAC comparatively to VKA are limited, conflicting, potentially biased and finally inconclusive in this population. Nevertheless, this population is the most at risk for nv AF and the population with the highest risk of both AF-related thrombotic events and anticoagulant-related major bleedings.

* Objectives: The aim of the study is to assess and compare the real benefits and harms of the two therapeutic strategies available in routine practice, for the anticoagulation in patients 75 years old or more suffering from nvAF. The main objective is to estimate and compare DOAC and VKA in terms of major bleeding, thrombotic events (TE) and death of all cause in 75 years old or more suffering from nv AF. The secondary objectives are to identify factors associated with the occurrence of these events, taking into account the type of anticoagulant, to identify factors associated with the occurrence of these events, taking into account switches from VKA to DOAC or DOAC to VKA, and to describe the utilization patterns of oral anticoagulants.
* Design and statistical analyses: An observational study will be conducted in the French administrative database (SNIIRAM). The SNIIRAM database contains anonymous and prospectively recorded data about all beneficiaries' medical reimbursements including age, gender, long-term chronic disease (LTD), date of death, all out-hospital health-spending reimbursements and all patients' hospitalizations. We will include all octo+ patients they care for, newly treated ("new users") with an oral anticoagulant (VKA or DOAC) for nv AF, at the date of first prescription of oral anticoagulant. From the date, patients data will be collected during at least 2 years. To assess the principal endpoint, we will estimate the time between the date of inclusion and the date of occurrence of a major thromboembolic event, major bleeding event, or death from any cause, whichever comes first. Exposure will be considered as time-dependant. The total number of patients expected is 150 000."

ELIGIBILITY:
Inclusion Criteria:

* Beneficiaries initiating a treatment by VKA or NOAC during the inclusion period (July 1, 2011 to December 31, 2014).
* Aged ≥ 75 years old et the time of OAC initiation.
* Presenting with an non valvular atrial fibrillation (nv AF).

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Beneficiaries aged ≥ 75 years old initiating a treatment by VKA or NOAC with an non vavular atrial fibrillation (nv AF).
Sampling Method: Non-Probability Sample
Enrollment: 150000 (Estimated)
Dates: Start 2016-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Composite of major thromboembolic events, major bleeding events or death from any cause | 2 years
  Major thromboembolic events include: Ischemic stroke, systemic or pulmonary embolism. Major bleeding is defined as a bleeding resulting in death or requiring hospital admission

SECONDARY OUTCOMES:
Potential risk factors for major bleeding and TE events in patients exposed to oral anticoagulant | 1 year
Patterns of use of OAC | 1 year
  Patterns of use will be described by : characteristics of the treated population (age, comorbidities leading to hospitalization), drug dose and regimen, time on treatment, concomitant drugs

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Bonnet-Zamponi, MD, Principal Investigator — Assistance Publique Hopitaux de Paris

IPD SHARING:
Plan to Share IPD: Undecided